CLINICAL TRIAL: NCT03110835
Title: Use of Low-dose Radioiodine for Ablation of Thyroid Remnants in Patients With Graves' Disease Following Thyroidectomy
Brief Title: Low-dose Radioiodine Ablation in Graves' Disease
Acronym: LORIGRAVES
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Other Study IDs: LORIGRAVES
Record Dates: First submitted 2017-03-14; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Diseases
MeSH Terms: conditions — Thyroid Diseases | interventions — Iodine-131

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 15 mCi radioiodine: 6 patients with low risk differentiated thyroid cancer, as determined by histology
  Interventions: Radiation: Radioiodine
- 30 mCi radioiodine: 6 patients with low risk differentiated thyroid cancer, as determined by histology
  Interventions: Radiation: Radioiodine

INTERVENTIONS:
Radiation: Radioiodine — Administration of radioiodine
  Other Names: 131-Iodine

SUMMARY:
Graves' orbitopathy (GO) is an autoimmune condition almost always associated with autoimmune thyroid disease, especially Graves' disease (GD). According to the most widely accepted model, the autoantigen/s responsible for GO would include molecules expressed by thyroid epithelial cells that are present also in orbital tissues. The high likelihood that the etiologies of GO and of the underlying autoimmune thyroid diseases are somehow linked is confirmed by the very close relationship between GO, the onset and the course of Graves' diseases, the size of the thyroid gland, and most importantly, thyroid function and thyroid treatment. Based on these considerations, it has been proposed that complete removal of thyroid antigens and of thyroid infiltrating lymphocytes, the so called total thyroid ablation (TTA), may be followed by an attenuation of the immune reaction against orbital antigens, and ultimately by an amelioration of GO. The possibility that TTA, achieved by near total thyroidectomy followed by radioiodine, may be beneficial for GO was initially suggested by two retrospective studies and more recently by two prospective, randomized clinical trials conducted in patients with moderate GO treated with intravenous glucocorticoids. Although there seemed to be no difference in the long term, compared with near total thyroidectomy alone TTA was associated with a shorter time required for GO to improve, or anyway to reach its best possible outcome, and with a lesser requirement for additional treatments in order for GO to improve.

TTA is usually performed with a radioiodine dose of 30 millicurie (mCi), administered after 2 injections of recombinant human thyrotropin TSH (rhTSH), the latter in order to induce radioiodine uptake by thyroid remnants. According to the Italian legislation the administration of such a dose of radioiodine must be followed by a 24 hours protected hospitalization. Clearly, this necessity implies a remarkable increase of the waiting list, due to the limited number of radiation-isolated beds available and, concerning GO patients, to the competition with patients with thyroid cancer. In contrast, a radioiodine dose of 15 mCi can be performed in out-patients without hospitalization and with much lower costs. Concerning GD patients, they usually have serum TSH-receptor stimulating antibodies that ay persist after thyroidectomy and that may increase radioiodine uptake along with rhTSH, possibly resulting in the need for a lower dose of radioiodine to ablate thyroid remnants. In order to investigate whether this is the case, the present study was designed in patients with GD. The study design was to include patients scheduled to radioiodine treatment with 30 or 15 mCi after administration of rhTSH, being the primary outcome the values of serum thyroglobulin at peak after administration of rhTSH 6 months after radioiodine, as a measure of the presence of residual thyroid tissue.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease at histology
* Thyroid cancer at histology
* Undetectable serum anti-thyroglobulin autoantibodies
* Informed consent

Exclusion Criteria:

* Detectable serum anti-thyroglobulin autoantibodies
* lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thyroidectomized patients with Graves' hyperthyroidism and GO undergoing radioiodine ablation with either 15 or 30 mCi of 131I
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
rhTSH-stimulated serum thyroglobulin (Tg) at 6 months | 6 months
  Measurement of Tg after 2 injections of rhTSH

SECONDARY OUTCOMES:
Serum Tg | 6 months
  Measurement of Tg prior to injections of rhTSH

IPD SHARING:
Plan to Share IPD: No